CLINICAL TRIAL: NCT00944333
Title: Second Generation" Drug-Eluting Stents Implantation Followed by Six Versus Twelve-Month - Dual Antiplatelet Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: STOP due to recent data in literature questioning the need to continue DAP beyond six months in patients with stable coronary artery stenting with DES.
Sponsor: Fondazione Evidence per Attività e Ricerche Cardiovascolari ONLUS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Security
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Angina Pectoris; Silent Ischemia
Keywords: second generation DES; clopidogrel; dual platelet therapy; patients with documented silent ischemia; unstable angina pectoris (Braunwald Classification); Diagnosis of angina pectoris (CCS)
MeSH Terms: conditions — Angina Pectoris; Angina, Unstable | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel 6 (Experimental): 6 month dual antiplatelet therapies in patients after second generation DES implantation
  Interventions: Drug: Clopidogrel
- Clopidogrel 12 (Experimental): 12 month dual antiplatelet therapies in patients after second generation DES implantation
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — 300-600 loading dose 75 mg/die for 6 months
  Arms: Clopidogrel 6
Drug: Clopidogrel — 300-600 loading dose 75 mg/die for 12 months
  Arms: Clopidogrel 12

SUMMARY:
Prospective, randomized, non-inferiority, multicenter, international study.In total 4000 patients (70 centers in Europe) with de novo lesions in native coronary arteries who meet the eligibility criteria randomized to 6 versus 12 month dual antiplatelet therapies following a second generation DES implantation.

Assuming that the true proportion of thrombotic events is equal to 2.3% for both regimens (6-month and 12-month clopidogrel) 2000 patients for each treatment group are necessary to demonstrate a non-inferiority of the 6-months regimen if the proportion of thrombotic events will be no more than 3.5% with a power of 0.80 and a significance level of 0.05 (one-tail).

If the non-inferiority hypothesis will be rejected, the superiority hypothesis (12-months regimen is superior to the 6-months-regimen) will be tested at a significance level of 0.05 (two-tails).

The maximal not clinically relevant difference for the non-inferiority hypothesis of 1.2 % more thrombotic events has to be considered together with the lower expected number of bleeding events in the 6-months regimen.

All the analysis will be done as "intention-to-treat" analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I,II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II-III) OR patients with documented silent ischemia, all treated with a second generation drug eluting stent
* Presence of one or more de novo stenosis equal or greater than 70% in a native coronary artery, treated with a Resolute drug eluting stent
* Patient is > 18 years of age (or minimum age as required by local regulations).
* The patient has consented to participate by signing the "Patient Informed Consent Form""
* The patient is willing and able to cooperate with study procedures and required follow up visits
* Any type of lesion or number of lesion can be included in this trial unless specifically detailed in the exclusion criteria.
* At least one second generation DES implanted in the target lesion in the last 24 hours
* No other DES implanted before the target procedure
* No BMS implanted in the 12 months before the target procedure

Exclusion Criteria:

* Patients treated for lesions in venous or arterial grafts
* Patients treated for in-stent restenosis
* Patients treated for Unprotected Left Main lesions
* ST elevation myocardial infarction in the 48 hours prior to the procedure
* Non ST elevation myocardial infarction
* Patients with LVEF≤30%
* Women with known pregnancy or who are lactating
* Patients with hypersensitivity or allergies to hepari, or any other analogue or derivative, cobalt, chromium, nickel, molybdenum or contrast media.
* Patients with chronic renal insufficiency
* Contraindication to the use of clopidogrel and/or ASA:

  * History of drug allergy to thienopyridine derivatives or ASA
  * History of clinically significant or persistent thrombocytopenia or neutropenia
  * Active bleeding or significant risk of bleeding, such as elderly patients receining fibrinolytic therapy and other potent antithrombotic agents, severe hepatic insufficiency, current peptic ulceration, proliferative diabetic retinopathy
  * Uncontrolled hypertension
* Current medical condition with a life expectancy of less than 24 months.
* The subject is participating in another device or drug study
* Subject must have completed the follow-up phase of any previous study at least 30 days prior to enrolment in this trial.
* Patients with medical conditions that preclude the follow-up as defined in the protocol or that otherwise limits participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1378 (Actual)
Dates: Start 2009-07; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Definite and/or probable stent thrombosis occurring between 6 and 24 months | 24 months

SECONDARY OUTCOMES:
Composite of major adverse cardiac events (MACE) defined as the occurrence at 24 months of cardiac death, or myocardial infarction, or urgent target vessel revascularization (cardiac bypass surgery, or repeat PTCA) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Fondazione Centro S. Raffaele Del Monte Tabor -, Milano (mi), Italy

REFERENCES:
- [Derived] Colombo A, Chieffo A, Frasheri A, Garbo R, Masotti-Centol M, Salvatella N, Oteo Dominguez JF, Steffanon L, Tarantini G, Presbitero P, Menozzi A, Pucci E, Mauri J, Cesana BM, Giustino G, Sardella G. Second-generation drug-eluting stent implantation followed by 6- versus 12-month dual antiplatelet therapy: the SECURITY randomized clinical trial. J Am Coll Cardiol. 2014 Nov 18-25;64(20):2086-97. doi: 10.1016/j.jacc.2014.09.008. Epub 2014 Sep 15. PMID 25236346